CLINICAL TRIAL: NCT02965898
Title: The Effect of Vitamin D Substitution on Pancreatic Parenchyma and Development of Fibrosis After First Acute Alcoholic Pancreatitis: A Randomized Prospective Trial
Brief Title: The Effect of Vitamin D Substitution on the Development of Chronic Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Principal Investigator, Mikael Parhiala, PhD canditate, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R16004
Record Dates: First submitted 2016-09-23; First posted 2016-11-17 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pancreatitis
Keywords: chronic pancreatitis; vitamin d; pancreatitis; Pancreatic stellate cell; rct
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Vitamin D 100ug (Active Comparator): The highest safest dose. Expected to lower risk of chronic pancreatitis after acute pancreatitis.
  Interventions: Dietary Supplement: Vitamin D 100ug
- Vitamin D 10ug (Placebo Comparator): Placebo dose. Minimal recommended dose
  Interventions: Dietary Supplement: Vitamin D 10ug

INTERVENTIONS:
Dietary Supplement: Vitamin D 100ug — Vitamin D 100 ug from Orion Pharma. Safest highest daily dose of vitamin D.
  Arms: Vitamin D 100ug
Dietary Supplement: Vitamin D 10ug — Placebo dose. Minimal recommended dose.
  Arms: Vitamin D 10ug

SUMMARY:
Acute pancreatitis (AP) may develop to chronic pancreatitis (CP). In Finland, the ethiology is alcohol in about 80% of the cases. Several symptoms lower the quality of life in CP patients, including abdominal pain, exocrine and endocrine pancreatic insufficiency.

Recently, the investigators and others have found that vitamin D may protect from the formation of fibrosis on cellular level. The investigators hypothesized that after the first AP they may be able to protect the formation of fibrosis leading to CP with Vitamin D, and designed this RCT.

The aim is to study whether the investigators can prevent CP with vitamin D substitute.

In this randomized controlled patient study, the patients after their first AP are randomized to have either a normal recommended (10 μ) or a largest safe dose (100 μg). of vitamin D substitute daily. The patients are examined by MRI/MRCP imaging and laboratory tests at the baseline after recovery from AP and yearly then after.

Primary endpoint is the development of parenchymal changes possibly related to fibrosis. Secondary endpoints are the development of CP with Mannheim criteria, CP related complications and mortality.

The first analysis will be done after 7 years.

The enrollment will begin 26.9.2016

ELIGIBILITY:
Inclusion Criteria:

* First alcohol induced acute pancreatitis
* Willing to participate in a 3 year RCT

Exclusion Criteria:

* Renal failure
* Hypercalcemia
* High serum levels of vitamin D
* Unwilling to participate

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
The development of parenchymal changes possibly related to fibrosis after acute pancreatitis analysed by magnetic resonance cholangiopancreatography imaging texture analysis | 3 years
  A radiologist analyses the pancreatic parenchymal changes from MRCP images

SECONDARY OUTCOMES:
The development of chronic pancreatitis (CP) with Mannheim criteria | 3 years
  The diagnostic Mannheim criteria include laboratory tests for measuring the endocrine and exocrine function of the pancreas and MRI/MRCP for measuring pancreatic duct lesions and calcifications.
The development of complications related to chronic pancreatitis | 3 years
  The complications are registered from the participants medical records.
Mortality related to chronic pancreatitis | 3 years
  The mortality is registered from the participants medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Yes
The data will be written into an article, which shall be displayed in a national and international forum.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Sherman MH, Yu RT, Engle DD, Ding N, Atkins AR, Tiriac H, Collisson EA, Connor F, Van Dyke T, Kozlov S, Martin P, Tseng TW, Dawson DW, Donahue TR, Masamune A, Shimosegawa T, Apte MV, Wilson JS, Ng B, Lau SL, Gunton JE, Wahl GM, Hunter T, Drebin JA, O'Dwyer PJ, Liddle C, Tuveson DA, Downes M, Evans RM. Vitamin D receptor-mediated stromal reprogramming suppresses pancreatitis and enhances pancreatic cancer therapy. Cell. 2014 Sep 25;159(1):80-93. doi: 10.1016/j.cell.2014.08.007. PMID 25259922
- [Background] Blauer M, Sand J, Laukkarinen J. Physiological and clinically attainable concentrations of 1,25-dihydroxyvitamin D3 suppress proliferation and extracellular matrix protein expression in mouse pancreatic stellate cells. Pancreatology. 2015 Jul-Aug;15(4):366-71. doi: 10.1016/j.pan.2015.05.044. Epub 2015 May 14. PMID 26005021
- [Background] Hathcock JN, Shao A, Vieth R, Heaney R. Risk assessment for vitamin D. Am J Clin Nutr. 2007 Jan;85(1):6-18. doi: 10.1093/ajcn/85.1.6. PMID 17209171
- [Background] Steffensen LH, Jorgensen L, Straume B, Mellgren SI, Kampman MT. Can vitamin D supplementation prevent bone loss in persons with MS? A placebo-controlled trial. J Neurol. 2011 Sep;258(9):1624-31. doi: 10.1007/s00415-011-5980-6. Epub 2011 Mar 13. PMID 21400196
- [Background] Stallings VA, Schall JI, Hediger ML, Zemel BS, Tuluc F, Dougherty KA, Samuel JL, Rutstein RM. High-dose vitamin D3 supplementation in children and young adults with HIV: a randomized, placebo-controlled trial. Pediatr Infect Dis J. 2015 Feb;34(2):e32-40. doi: 10.1097/INF.0000000000000483. PMID 24988118
- [Derived] Parhiala M, Aronen A, Ukkonen M, Haukijarvi E, Pappinen P, Rinta-Kiikka I, Laukkarinen J. High-Dose Vitamin D and Early Chronic Pancreatitis-Related Changes After Acute Pancreatitis: A Randomized Dose Controlled Trial. Dig Dis Sci. 2026 Jan 26. doi: 10.1007/s10620-026-09688-x. Online ahead of print. PMID 41588283